CLINICAL TRIAL: NCT06488235
Title: Evaluation Qualitative de Programmes d'Education Thérapeutique d'obésité pédiatrique
Brief Title: Qualitative Evaluation of Pediatric Obesity Therapeutic Education Programs
Acronym: QUALIPOP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 23_0304
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Obesity
Keywords: pediatric obesity; attrition; Educational care program
MeSH Terms: conditions — Pediatric Obesity; Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obese adolescents over 12 years of age and their parents: Children who have started an educational care program between 2017 and 2022 at one of the four participating centers and have stopped the educational care program early.
  Child over 12 years of age at the time of the focus group.

SUMMARY:
Obesity concerns almost the entire planet and is considered in France as a major public health issue: 17% of children are overweight and 4% obese.

Because of this situation, the public authorities have set up programs in order to overcome obesity. Accompanying the child and its family in a process of change through Educational care program seems to be the most suitable. Unfortunately, the abandonment rate of these programs is often high.

DETAILED DESCRIPTION:
The main aim of this study is to explore, describe and understand the phenomenon of attrition in different pediatric obesity Educational care program since 2017 by collecting their experience by describing and characterizing the reasons for attrition reported by the patients included.

ELIGIBILITY:
Inclusion Criteria:

* Children who have started an educational care program between 2017 and 2022 at one of the four participating centers.
* Children whose parents or legal guardians have signed the program participation letter.
* Children who have participated in at least one group session and have stopped the educational care program early.
* Children whose parents have agreed to take part in the focus group for themselves and their child.
* Children over 12 years of age at the time of the focus group.

Exclusion Criteria:

* Child who has completed the Educational Care program
* Parent/child pairs where at least 1 of the 2 refused to take part in the study

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents who have stopped their Educational Care Programme (early in 1 of the 4 centers over the last 3 years.
  They may still be receiving individual follow-up at their center, or may have had a break in care.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Categorization of the reasons given by children and parents | during the data analysis, either 6 months following the focus group period
  Description and categorization of the reasons given by children and parents

SECONDARY OUTCOMES:
Mirroring of the respective experiences of attrition by children | during the data analysis, either 6 months following the focus group period
  Description and mirroring of the respective experiences of attrition by children

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Labarre, Principal Investigator — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No